CLINICAL TRIAL: NCT01703169
Title: Efficacy and Safety of Eltrombopag In Patients With Severe and Very Severe Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI54443; ELT115895 (Other: Novartis)
Record Dates: First submitted 2012-09-27; First posted 2012-10-10 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Severe Aplastic Anemia; Very Severe Aplastic Anemia; Moderate Aplastic Anemia
Keywords: severe aplastic anemia; very severe aplastic anemia; moderate aplastic anemia; bleeding
MeSH Terms: conditions — Anemia, Aplastic; Hemorrhage | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eltrombopag (Experimental): Single arm study. Dose Escalation.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Oral eltrombopag 150mg/day by mouth starting on Day 1 with dose modification over 12 weeks to a maximum of 300mg/day determined by platelet count

SUMMARY:
The investigators hypothesis is that eltrombopag given to patients with moderate to very severe aplastic anemia will result in an increase in platelet counts. The investigators hypothesize that in patients with moderate to very severe aplastic anemia, treatment with eltrombopag will lead to fewer platelet transfusions, red blood cell transfusions, and fewer bleeding events. The investigators hypothesize that in patients with moderate to very severe aplastic anemia, eltrombopag will have an acceptable toxicity rate <3%, at doses that result in increased platelet counts. Finally the investigators hypothesize that plasma eltrombopag levels in peripheral blood will correlate with improved platelet counts.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent and any other authorizations required by local law (e.g., Protected Health Information [PHI])
* Have severe or very severe aplastic anemia, or moderate aplastic anemia with platelet counts that have dropped below 20,000/μl
* Have moderate, severe, or very severe aplastic anemia with moderate bleeding during or after a surgical procedure, (including bone marrow biopsy, lumbar puncture, thoracentesis, paracentesis, port placement, dermal biopsy) or minimal mucocutaneous bleeding otherwise noted
* Subjects with current or previous exposure to approved medications for the treatment of aplastic anemia will not be excluded; these include but may not be limited to, anti-thymocyte globulin (ATG), cyclosporine, corticosteroids, and G-CSF.

Exclusion Criteria:

* Have diagnosis of Fanconi anemia
* Have infection not adequately responding to appropriate therapy
* Have Paroxysmal Nocturnal Hemoglobinuria (PNH) clone size in neutrophils of greater than or equal to 50%
* Have known HIV positivity
* Have creatinine and/or blood urea nitrogen (BUN) ≥2 times the upper limit of normal
* Have serum bilirubin ≥ 1.5 times the upper limit of normal, or ≥4.0 times the upper limit of normal if the patient has been treated with ATG within three weeks of screening.
* Have AST and/or ALT ≥ 3 times the upper limit of normal
* Have hypersensitivity to eltrombopag or its components
* Have chemotherapy given less than or equal to 14 days prior to initiating the study medication. This does not include immunosuppressive agents and growth factor as described above
* Are female and are nursing or pregnant or are unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential
* Are unable to understand the investigational nature of the study or give informed consent
* Have a history of arterial or venous thrombosis within the last 1 year (excluding those due to indwelling lines)
* Have an ECOG performance status of 3 or greater
* Have had treatment with Campath within 6 months of entry into the study
* Have pre-existing cardiovascular disease (congestive heart failure with New York Heart Association [NYHA] grade III/IV), arrhythmia known to increase the risk of thromboembolic events (e.g. atrial fibrillation), unstable angina, or QTc > 450 msec (QTc 480 msec for subjects with bundle branch block), or myocardial infarction within the preceding 6 months) at study entry
* Have had other TPO-R agonists medication in the previous 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George M Rodgers, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eltrombopag
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eltrombopag
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: Count of Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Platelet Response
Description: Defined as a stable platelet count of 50,000/μl or more during any 4 week period within the possible 12 weeks while on study,and including maximal platelet counts achieved in patients with moderate to very severe aplastic anemia.
Time Frame: up to 12 weeks
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 13
proportion of participants | 0.23 [0.05 to 0.54]
Statistical Analysis 1: Comparison: Eltrombopag; Test type: Other; The proportion of platelet response in a previous study (PMID:22762314) was 0.36 (9/25). The null hypothesis of no difference between the platelet response rate in this study and that of the previous study was tested using a two-sided exact test of binomial proportions. A p-value of 0.40 was obtained. The threshold for significance was 0.05

2. Secondary Outcome: Platelet Count Twice Baseline.
Description: Proportion of subjects who achieve platelet counts at least twice their baseline value at any point while on study medication, in patients with moderate to very severe aplastic anemia.
Time Frame: Between weeks 1-12.
Population: Data was not collected for this outcome variable.
Arm/Group | Eltrombopag
Number analyzed (Participants) | 0

3. Secondary Outcome: Hematology Labs
Description: Association between eltrombopag use and response in hemoglobin, hematocrit, total white blood cell count, and absolute neutrophil count to be evaluate by maximal hemoglobin, hematocrit, total white blood cell count, and absolute neutrophil counts achieved in patients with moderate to very severe aplastic anemia
Time Frame: 12 weeks
Population: Data was not collected for this outcome variable.
Arm/Group | Eltrombopag
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Patients With AE to Measure Toxicity, Using NCI CTCAE
Description: Evaluated weekly, up to 12 weeks. Association between eltrombopag use, dose, and tolerability in patients with moderate to very severe aplastic anemia
Time Frame: 12 weeks
Population: Data was not collected for this outcome variable.
Arm/Group | Eltrombopag
Number analyzed (Participants) | 0

5. Secondary Outcome: Characterization of the PK Profile of Eltrombopag in Patients With Moderate to Very Severe Aplastic Anemia. Evaluated With AUC, Cmax, Cmin, Tmax.
Description: Samples will for PK analysis will collected as a trough level weeks 2, 6 and 12, prior to dose of eltrombopag. Additional PK level drawn at 2, 4 and 6 hours post-dose at the scheduled week 2 visit.
Time Frame: Weeks 2, 6 and 12
Population: Data was not collected for this outcome variable.
Arm/Group | Eltrombopag
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Approximately 3 years.
Arm/Group | Eltrombopag
All-Cause Mortality (participants affected / at risk) | 2/13
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eltrombopag (N=13)
congestive heart failure (Cardiac disorders) | 1 (1)
cholecystitis (Hepatobiliary disorders) | 1 (1)
syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eltrombopag (N=13)
abdominal pain (Gastrointestinal disorders) | 1 (2)
aches/pains (General disorders) | 2 (2)
anemia (Blood and lymphatic system disorders) | 3 (13)
anxiety (Psychiatric disorders) | 1 (1)
arrhythmia (Cardiac disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
purpura (Skin and subcutaneous tissue disorders) | 5 (8)
bronzing of the skin (Skin and subcutaneous tissue disorders) | 2 (3)
bruising (Injury, poisoning and procedural complications) | 3 (5)
chest pain (Cardiac disorders) | 1 (2)
chills (General disorders) | 1 (1)
confusion (Psychiatric disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
cramps (Musculoskeletal and connective tissue disorders) | 2 (2)
decreased lymphocyte count (Investigations) | 3 (22)
decreased neutrophil count (Investigations) | 3 (17)
thrombocytopenia (Investigations) | 6 (24)
dehydration (Metabolism and nutrition disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (4)
dizziness (Nervous system disorders) | 1 (1)
dry mouth (Gastrointestinal disorders) | 1 (1)
dry skin (Skin and subcutaneous tissue disorders) | 1 (3)
dysgeusia (Nervous system disorders) | 2 (3)
dysuria (Renal and urinary disorders) | 1 (1)
ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2)
edema (General disorders) | 4 (10)
Alkaline phosphatase increased (Investigations) | 1 (1)
elevated ALT (Investigations) | 3 (10)
elevated AST (Investigations) | 3 (5)
elevated bilirubin (Investigations) | 4 (7)
elevated creatinine (Investigations) | 3 (8)
hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
erythema (Skin and subcutaneous tissue disorders) | 1 (1)
fatigue (General disorders) | 7 (8)
gum hypertrophy (Infections and infestations) | 1 (1)
gum lesions (Infections and infestations) | 1 (1)
facial hair growth (Skin and subcutaneous tissue disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
hematoma (Vascular disorders) | 1 (1)
hot flashes (Vascular disorders) | 1 (1)
hypertension (Vascular disorders) | 2 (2)
hypoalbunemia (Investigations) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 2 (5)
hyponatremia (Metabolism and nutrition disorders) | 2 (5)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
insomnia (Psychiatric disorders) | 2 (2)
jaundice (Skin and subcutaneous tissue disorders) | 2 (2)
menorrhagia (Reproductive system and breast disorders) | 2 (3)
mouth sores (Skin and subcutaneous tissue disorders) | 2 (2)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
otitis externa (Infections and infestations) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (3)
night sweats (General disorders) | 1 (1)
opacity (Eye disorders) | 1 (1)
pain (General disorders) | 5 (7)
pallor (Skin and subcutaneous tissue disorders) | 3 (3)
petechiae (Blood and lymphatic system disorders) | 11 (18)
port leak (General disorders) | 1 (1)
pyelonephritis (Renal and urinary disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 3 (4)
rectal hemorrhage (Gastrointestinal disorders) | 1 (2)
renal insufficiency (Renal and urinary disorders) | 2 (2)
respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sciatica (Nervous system disorders) | 1 (1)
scleral icterus (Eye disorders) | 2 (2)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
spelnomegaly (Hepatobiliary disorders) | 1 (1)
thrush (Skin and subcutaneous tissue disorders) | 1 (1)
transfusion reaction (Blood and lymphatic system disorders) | 1 (1)
tremor (Nervous system disorders) | 1 (1)
urinary tract infection (Infections and infestations) | 2 (3)
weight gain (Investigations) | 4 (4)

LIMITATIONS AND CAVEATS:
Certain data regarding the primary outcome and adverse events were inadvertently not captured during the clinical investigation resulting in insufficient data for statistical analysis and publication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes